CLINICAL TRIAL: NCT03851081
Title: A Multi-Center, Open-Label Phase 1b/2 Study of Inotuzumab Ozogamicin and Vincristine Sulfate Liposome in Adult Patients With Relapsed/Refractory B Lineage Acute Lymphoblastic Leukemia (B-ALL)
Brief Title: Inotuzumab Ozogamicin and Vincristine Sulfate Liposome in Treating Patients With Relapsed or Refractory CD22+ B-cell Acute Lymphoblastic Leukemia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 66818; NCI-2019-00565 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 66818 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-02-19; First posted 2019-02-22 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation Recipient; Blasts 5 Percent or More of Bone Marrow Nucleated Cells; Blasts 5 Percent or More of Peripheral Blood White Cells; CD22 Positive; Lymphoblasts 20 Percent or More of Bone Marrow Nucleated Cells; Lymphoblasts 20 Percent or More of Peripheral Blood White Cells; Recurrent B Acute Lymphoblastic Leukemia; Refractory B Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma | interventions — Inotuzumab Ozogamicin; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (inotuzumab ozogamicin, liposomal vincristine) (Experimental): See Detailed Description.
  Interventions: Biological: Inotuzumab Ozogamicin; Other: Quality-of-Life Assessment; Drug: Vincristine Sulfate Liposome

INTERVENTIONS:
Biological: Inotuzumab Ozogamicin — Given IV
  Other Names: Besponsa; CMC-544; Way 207294; WAY-207294
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Vincristine Sulfate Liposome — Given IV
  Other Names: Marqibo

SUMMARY:
This phase Ib/II trial studies side effects and best dose of inotuzumab ozogamicin and how well it works when given together with vincristine sulfate liposome in treating patients with CD22 positive (+) B-cell acute lymphoblastic leukemia that has come back or dose not respond to treatment. Inotuzumab ozogamicin is a monoclonal antibody, called inotuzumab, linked to a toxic agent called ozogamicin. Inotuzumab attaches to CD22+ cancer cells in a targeted way and delivers ozogamicin to kill them. Drugs used in chemotherapy, such as vincristine sulfate liposome, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving inotuzumab ozogamicin and vincristine sulfate liposome together may work better in treating patients with CD22+ B-cell acute lymphoblastic leukemia compared to giving inotuzumab ozogamicin or vincristine sulfate liposome alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of vincristine sulfate liposome (liposomal vincristine) and inotuzumab ozogamicin combination therapy in adult patients with relapsed and/or refractory B lineage acute lymphoblastic leukemia (B-ALL).

II. To evaluate the overall response rate (ORR consisting of complete remission [CR], morphologic CR with incomplete blood count recovery [CRi], of combination therapy with liposomal vincristine and inotuzumab ozogamicin in adult patients with relapsed and/or refractory B lineage acute lymphoblastic leukemia.

SECONDARY OBJECTIVES:

I. To evaluate the leukemia-free survival (LFS) and overall survival (OS) of patients treated with this combination.

II. To evaluate the number of patients able to proceed onto subsequent hematopoietic stem cell transplantation (HSCT) following combination therapy following combination therapy.

III. To evaluate the overall incidence of unique toxicities associated with these agents, specifically peripheral neuropathy following vincristine sulfate liposome and veno-occlusive disease of the liver (VOD) following inotuzumab ozogamicin therapy.

EXPLORATORY OBJECTIVES:

I. To explore minimal residual disease (MRD) as a potential correlative biomarker of response to combination vincristine sulfate liposome and inotuzumab ozogamicin therapy.

II. To explore potential biomarkers of response to vincristine sulfate liposome and inotuzumab ozogamicin therapy.

III. To perform an analysis of the estimated cost of outpatient administration of vincristine sulfate liposome and inotuzumab ozogamicin.

IV. To evaluate quality of life (QOL) of patients with relapsed/refractory B-ALL treated with vincristine sulfate liposome and inotuzumab ozogamicin.

OUTLINE: This is a phase Ib, dose-escalation study of inotuzumab ozogamicin followed by a phase II study.

INDUCTION/RE-INDUCTION: Patients receive vincristine sulfate liposome intravenously (IV) over 1 hour and inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 2 cycles in the absence of disease progression or unacceptable toxicity. Patients who achieve clinical benefit, defined as stable disease (SD), PR or CR, or CRi after 1-2 cycles, will continue on to maintenance therapy for up to 4-5 cycles. Patients who do not achieve clinical benefit after cycle 1 but do not experience dose-limiting toxicities (DLTs) receive a second cycle of vincristine sulfate liposome and inotuzumab ozogamicin.

MAINTENANCE: Patients receive vincristine sulfate liposome IV over 1 hour on days 1 and 15 and inotuzumab ozogamicin IV over 1 hour on days 1, 8, and 15. Treatment repeats every 28 days for up to 4-5 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group performance status between 0-2
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance (Cockcroft and Gault) > 30 mL/min
* Alanine aminotransferase (ALT) =< 5 x ULN
* Total bilirubin= < 1.5 x ULN
* Left ventricular ejection fraction (LVEF) >= 40% as assessed by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scan performed within 28 days of enrollment
* Diagnosis of relapsed/refractory CD22+ B-cell ALL with disease in the bone marrow and/or peripheral blood by morphology (>=5% blasts). CD22-positive B-ALL is defined as expression by at least 20% of malignant lymphoblasts as determined by local flow cytometry and/or immunohistochemistry from a peripheral blood and/or bone marrow sample obtained within 2 weeks of screening
* Relapsed or refractory disease, defined as second or greater bone marrow relapse from CR or overall response or, disease has progressed following two or more anti-leukemia therapies. Specifically:

  * Any bone marrow relapse after allogeneic HSCT: subjects must be at least 1 month from HSCT at the time of screening and off immunosuppressive medication for at least 2 weeks at time of initial treatment (with the exception of low-dose steroids =< 20 mg prednisone equivalent) and have no active graft versus (vs.) host disease (GVHD);
  * Philadelphia chromosome (Ph) negative B-ALL which has not achieved CR or CRi after at least 2 attempts at remission induction using standard intensive chemotherapy regimen(s);
  * Philadelphia chromosome (Ph) positive B-cell ALL intolerant to or ineligible for BCR-ABL tyrosine kinase inhibitor (TKI) therapy or with disease which has progressed after at least two lines of prior TKI therapy
* Participants of childbearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry and for females, at least 8 months after the final dose of inotuzumab ozogamicin. Males with female partners of childbearing potential must agree to use adequate contraceptive prior to study entry and for at least 5 months after the final dose of inotuzumab ozogamicin. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Receipt of chemotherapy, radiotherapy, or investigational drug therapy within 2 weeks prior to treatment on study or those who have not recovered from adverse events due to agents administered > 2 weeks earlier
* Participants on oral or injectable calcineurin inhibitors (e.g., cyclosporin, tacrolimus) within 4 weeks prior to study enrollment

  * Active central nervous system involvement; patients who have a history of central nervous system (CNS) disease which has been effectively treated (as defined by at least one negative cerebrospinal sample prior to screening) are eligible
* Prior malignancy, unless treated with curative intent and with no evidence of active disease present for > 5 years before screening, with the following exceptions:

  * Subjects with stage I breast cancer that has been completely and successfully treated, requiring no therapy or only anti-hormonal therapy
  * Subjects with T1N0M0 or T2N0M0 colorectal cancer who have been completely and successfully resected and who are disease-free for > 2 years prior to screening
  * Subjects with indolent prostate cancer, defined as clinical stage T1 or T2a, Gleason score =< 6, and prostate-specific antigen (PSA) < 10 ng/mL, requiring no therapy or only anti-hormonal therapy
  * Subjects with a history of basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix, fully resected, and with no evidence of active disease
* Uncontrolled intercurrent medical illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that in the opinion of the investigator would limit compliance with study requirements
* Uncontrolled systemic fungal, bacterial, viral, or other infection defined as exhibiting ongoing signs and symptoms due to infection despite appropriate anti-infective therapy at time of screening
* Pregnant or nursing female participants
* Known active hepatitis B, known active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of screening
* Presence of grade II-IV acute or extensive chronic graft versus host disease (GVHD) at time of screening
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug including, but not limited to, medical, psychological, familial, social, or geographical considerations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2023-01-21 (Estimated); Study Completion 2024-01-21 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) (Phase Ib) | Up to 28 days
  The maximum dose level will be reached when 1 or fewer DLTs are observed in 6 patients.
Overall response rate (ORR) (Phase II) | Up to 12 months after last dose of study treatment
  Defined as complete remission (CR), morphologic CR with incomplete blood count recovery (CRi), partial remission (PR), hematological improvement (HI) based on modified International Working Group (IWG) criteria. Response is treated as a dichotomous variable and will be summarized by dose level using frequencies and relative frequencies. The ORR will be estimated using an 80% confidence interval obtained by Jeffrey?s prior method.
Incidence of adverse events (AEs) | Up to 12 months after last dose of study treatment
  Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4 and defined as the number of patients who received study combination who developed subsequent vascular occlusive disease (VOD) or neurological toxicities. The observed AEs and DLTs will be summarized by dose level and grade using frequencies and relative frequencies. AE and DLT rates will be estimated with 90% confidence intervals obtained using Jeffrey?s prior method.

SECONDARY OUTCOMES:
Leukemia-free survival (LFS) | Time from enrollment until disease progression/recurrence, death due to any cause, or last follow-up, assessed up to 12 months after last dose of study treatment
  Will be based on modified IWG criteria. Will be summarized by dose level using standard Kaplan-Meier methods. Estimates of the median LFS will be obtained with 90% confidence intervals.
Overall survival | Time from enrollment until death due to any cause or last follow-up, assessed up to 12 months after last dose of study treatment
  Will be based on modified IWG criteria. Will be summarized by dose level using standard Kaplan-Meier methods. Estimates of the median OS will be obtained with 90% confidence intervals.
Number of patients who proceed onto subsequent hematopoietic stem cell transplantation (HSCT) | Up to 12 months after last dose of study treatment
  The post-therapy HSCT status will be summarized by dose level using frequencies and relative frequencies. The HSCT rate will be estimated with 90% confidence intervals obtained using Jeffrey?s prior method.
Number of patients who developed subsequent neurological toxicities and VOD | Up to 12 months after last dose of study treatment
  The VOD and neurological toxicities will be summarized by dose level using frequencies and relative frequencies. The toxicity rates will be estimated with 90% confidence intervals obtained using Jeffrey?s prior method.

OTHER OUTCOMES:
Minimal residual disease (MRD) after treatment | Up to 12 months after last dose of study treatment
Change in quality of life (QOL) | Baseline up to 6 months
  Will be analyzed using the Functional Assessment of Cancer Therapy - Leukemia (FACT-Leu).
Estimated cost analysis for administration of treatment | Up to 12 months after last dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eunice S Wang, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States